CLINICAL TRIAL: NCT04314869
Title: Feasibility Study of Uterus Transplantation Procedure From a Live Donor Obtaining the Graft by Laparoscopy
Brief Title: Uterus Transplantation Procedure From a Live Donor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Francisco Carmona, Head of Gynecology Department, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUX2020
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Rokitansky Kuster Hauser Syndrome; Sterility, Female
Keywords: minimally invasive surgery; uterus transplantation; living donor; absolut uterine factor
MeSH Terms: conditions — Mullerian aplasia; Infertility, Female | interventions — Embryo Transfer; Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recipient (Experimental): Patient with absolut uterine factor will undergo uterus transplantation.
  Interventions: Procedure: Uterus transplantation

INTERVENTIONS:
Procedure: Uterus transplantation — Patient will undergo surgery in order to transplant the graft (uterus). After that, a follow-up in order to detect early rejection. After 6 months, embryo transfer will be perfomed. Labour route will be C-Section. Two pregnancies are agreed, and after the second one, a hysterectomy will be performed in order to remove the graft.
  Other Names: Ovarian estimulation; Immunosupression treatment; Embryo transfer; C-section

SUMMARY:
Absolut uterine factor, meaning the absence of uterus, represents a cause for sterility without the possibility of a present treatment. The uterine factor affects millions of women and may be due to congenital problems, such as the Muller anomalies (Mayer Rockitansky Syndrome) or acquired by previous hysterectomy or intrauterine adhesions (Asherman's Syndrome). The uterine transplant would represent the only possibility for patients with an absolute uterine factor to achieve both genetic and gestational maternity.

DETAILED DESCRIPTION:
To obtain by laparoscopy a viable uterus for transplantation from a living donor is feasible. The laparoscopic procedure increases safety and provides the benefits of minimally invasive surgery to the grafting technique already described by laparotomy. The objective of the present study is to develop a pilot program in the transplant of a living donor. We include 5 pairs of uterine donor-transplant recipients indicated for sterility by absolute uterine factor due to Mayer Rokitansky Syndrome. Patients will undergo surgery for this transplant and after 6 months of it with correct function of the graft, embryos will be transferred in order to achieve pregnancy. C-section will be performed for delivery. The attempt of two gestations (if there are sufficient cryopreserved embryos for a second gestation) and withdrawing the graft (hysterectomy) and, therefore, immunosuppression is agreed.

ELIGIBILITY:
Inclusion Criteria Recipient:

* Patient with sterility for absolute uterine factor (malformation or previous surgery for benign processes).
* Age <40 years.
* Absence of pathology that contraindicates a complex surgical process, immunosuppression or gestation.
* Positive results to the IVF cycle prior to the surgery, obtaining quality embryos.
* Acceptance to participate in the study signing the informed consent.

Exclusion Criteria Recipient:

* Medical or surgical pathology that contraindicates a complex pelvic surgical procedure.
* Medical conditions that contraindicate, may aggravate or complicate the immunosuppressor treatment, such as neoplastic or preneoplasic diseases, chronic infectious diseases, autoimmune diseases, renal or liver failure.
* Medical or surgical pathology that contraindicates pregnancy.
* Anatomic alterations or vascular pathology that might difficult the vascular anastomosis: severe endometriosis, pelvic kidney, severe adherence syndrome or others.
* Uncontrolled psychopathology.

Inclusion Criteria donor:

* Age <65 years.
* First- or second-degree relatives.
* Completed reproductive desire.
* History of previous pregnancies and births.
* Absence of associated pathology that contraindicates prolonged and complex laparoscopic surgery (pneumopathies, heart disease, morbid obesity, …).
* Acceptance to participate in the study signing the informed consent

Exclusion Criteria donor:

* Potential future pregnancy desire.
* Surgery for the treatment of gender identity disorder.
* Infections: HIV or risk group, HBV-DNA and / or HBsAg positive, positive HCV, active bacterial sepsis, infections with multi-resistant bacteria, active tuberculosis or incomplete treatment of the same, Chagas disease, untreated active viral infections.
* Active malignant cancer of any location, except skin basal cell carcinoma. Treated cancer without current evidence of illness but with a follow-up of less than 5 years.
* Benign pelvic pathology: uterine fibroids, uterine malformations, severe endometriosis, severe adherence syndrome.
* Vascular pathology: malformations, atheromatosis, hypertensive or diabetic vasculopathy, connective tissue disease with vascular involvement.
* Premalignant pelvic pathology: pre-invasive cervical and/or vaginal, endometrial hyperplasia.
* BRCA mutation carriers or genes related to Lynch syndrome.
* History of implantation failure or multiple abortions of unknown cause.
* Contraindications for the surgical procedure of donation through laparoscopy: diabetes mellitus, liver disease, nephropathy, heart disease, pneumopathy, morbid obesity or high-risk cardiovascular factors.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It is a uterus transplantation program, it only includes women.
Enrollment: 10 (Estimated)
Dates: Start 2020-05-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of grafts obtained by laparoscopy | 2 years
  It is feasible to obtain the graft by laparoscopy

SECONDARY OUTCOMES:
Number of healthy newborns | 5 years
  A healthy newborn after C-section

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Carmona, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data, but we will publish all the results and protocols so other researchers have access to this information

REFERENCES:
- [Derived] Diaz-Feijoo B, Rius M, Gracia M, Musquera M, Magaldi M, Peri L, Alcaraz A, Carmona F. Donor robotic-assisted laparoscopy for uterus transplantation. Fertil Steril. 2022 Mar;117(3):651-652. doi: 10.1016/j.fertnstert.2021.11.026. Epub 2022 Jan 17. PMID 35058048